CLINICAL TRIAL: NCT00416533
Title: A Phase II Study of Taxotere (Docetaxel) Plus Adriamycin (Doxorubicin) and Prednisone (TAP) in Hormone-Refractory Prostate Cancer
Brief Title: Docetaxel, Doxorubicin, and Prednisone in Treating Patients With Advanced Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU-85302; CDR0000466318 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-BG04-264; AVENTIS-CCCWFU-85302
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Doxorubicin; Prednisone

INTERVENTIONS:
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: prednisone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, doxorubicin, and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel, doxorubicin, and prednisone together works in treating patients with advanced prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess prostate specific antigen response rate to docetaxel, doxorubicin hydrochloride, and prednisone in patients with hormone-refractory advanced prostate cancer.

Secondary

* Assess if treatment with docetaxel, doxorubicin hydrochloride, and prednisone will improve health-related quality of life of these patients.
* Assess the toxicity of docetaxel, doxorubicin hydrochloride, and prednisone.
* Assess response rate in measurable disease.

OUTLINE: Patients receive docetaxel IV over 1 hour on day 1, doxorubicin hydrochloride IV over 15 minutes on days 1 and 8, and oral prednisone once daily on days 1-21. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on day 1 of each course, after completion of 3 courses, and at disease progression.

After completing study treatment, patients are followed every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate with any of the following:

  * Prostate-specific antigen ≥ 10 mg/dL
  * Bone disease
  * Bidimensional soft tissue disease
  * Evaluable disease
* Advanced disease AND failed prior primary androgen ablation therapy, including anti-androgen withdrawal
* Disease not amenable to local curative treatment
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine < 2.0 mg/dL
* SGPT and SGOT < 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ ULN
* Hemoglobin ≥ 10 g/dL
* Ejection fraction ≥ 50%
* Peripheral neuropathy ≤ grade 1
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No previous history of or concurrent malignancy, except for any of the following:

  * Inactive nonmelanoma skin cancer
  * Disease-free for five or more years
  * Adequately treated stage I or II cancer from which patient is currently in complete remission
* No other serious medical illness that would limit survival to less than 3 months
* No psychiatric condition that would prevent informed consent
* No active, uncontrolled bacterial, viral, or fungal infection
* No hemorrhagic disorder
* No history of severe hypersensitivity reaction to other drugs formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No new hormonal treatment within the past 4 weeks
* No prior immunotherapy, chemotherapy, or bone-seeking radiopharmaceuticals (e.g., strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium)
* Prior bisphosphonates allowed
* At least 2 weeks since prior radiotherapy
* No other concurrent chemotherapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2004-08; Primary Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Torti, MD, MPH, Study Chair — Wake Forest University Health Sciences